CLINICAL TRIAL: NCT03939975
Title: A Prospective Study of Anti-PD-1 Inhibitors Therapy in Combination With Incomplete Thermal Ablation in Patients With Advanced Hepatocellular Carcinoma
Brief Title: Anti-PD-1therapy Combined With Thermal Ablation for Advanced HCC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Ming Zhao, Clinical Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2018-151-01
Record Dates: First submitted 2019-04-07; First posted 2019-05-07 (Actual); Last update posted 2019-08-19 (Actual); Status verified 2019-08

CONDITIONS: Carcinoma, Hepatocellular
Keywords: Hepatocellular carcinoma; Immunotherapy; Nivolumab; Pembrolizumab; Radiofrequency Ablation; Microwave ablation
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — pembrolizumab; Nivolumab

STUDY DESIGN:
Intervention Model Description: The study subjects were those who with advanced HCC that progressed on first-line sorafenib and treated with anti-PD-1 therapy in combination with incomplete thermal ablation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Study arm (Experimental): Patients with stable diseases or atypical progression to ICIs monotherapy would be additionally treated with incomplete thermal ablation along with ICIs therapy; and for those who with no lesions eligible for Incomplete ablation, ICIs would be given solely.
  Others with complete or partial responses would keep on going with mono-ICIs therapy.
  Interventions: Drug: pembrolizumab or nivolumab or JS001

INTERVENTIONS:
Drug: pembrolizumab or nivolumab or JS001 — ICIs therapy of nivolumab (3 mg/kg, per 2 weeks) or pembrolizumab (2 mg/kg, per 3 weeks) or JS001 (240mg, per 3 weeks) was performed until the off-treatment criteria were met. For participants with stable disease or atypical progression to ICIs therapy, thermal ablation of radiofrequency ablation or microwave ablation was performed addtionally.
  Other Names: computed tomography guided radiofrequency ablation; or computed tomography guided microwave ablation

SUMMARY:
The inhibition of programmed cell death protein 1 (PD-1) has shown promising antitumor activity in advanced hepatocellular carcinoma (HCC). Unfortunately, less than 20% of HCC have response. The effect of PD-1 blockade and incomplete thermal ablation in patients with advanced HCC is not yet clearly understood. This study aimed to analyze outcomes of advanced HCC treated with anti PD-1 inhibitors in combination with incomplete thermal ablation.

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) is ranked as the third leading cause of cancer death both worldwide and in the China. In the past decade, survivals of patients with advanced HCC or those who have progressed diseases following locoregional treatments can be increased with the multi-kinase inhibitor sorafenib, the first evidence identified drug for HCC. Recent clinical trials further verified some novel tyrosine kinase inhibitors such as regorafenib and cabozantinib, and two programmed cell death protein-1 (PD-1) immune checkpoint inhibitors (ICIs), nivolumab and pembrolizumab, as useful therapies in second line setting following sorafenib.

Advances in programmed cell death protein 1 (PD-1) blockade have shown an ORR of 15-17% and median survival time of 12.9-15.0 months among patients with advanced HCC. Of these, nivolumab and pembrolizumab have been accelerated approved as second-line treatment of advanced HCC. Notably, patients who have tumor responses maintain long-lasting disease control for 9.9-17months and still a large proportion of patients (81-83%) do not respond to mono PD-1 blockade, which emphasizing the need to explore strategies to increase the efficacy of immunotherapy.

An approach to expanding the benefit of ICIs may involve combinations with locoregional therapy like radiofrequency ablation (RFA) and transarterial chemoembolization (TACE), such treatments have been shown to boost tumor-specific T-cell response through release of TAAs from HCC cells. The intent-to-treat population of this study was a subset of patients receiving ongoing ICIs therapy for advanced HCC and is with stable disease or atypical responses in different lesions of the same individuals.

ELIGIBILITY:
Inclusion Criteria:

Eligible patients had pathological diagnosis of HCC by either surgical resection tissue or core needle biopsy; and had advanced stage of disease that is refractory to or is with unacceptable toxicity of sorafenib. Other eligibility criteria included: Child-Pugh A or B7 classification; Eastern Cooperative Oncology Group-performance status score 0-2; adequate bone marrow (leukocyte count >3.0 ×109/L, hemoglobin >8.0 g/L, and platelet count >60 ×109/L), liver (alanine aminotransferase and aspartate aminotransferase <200 IU/mL), renal (creatinine <1.5 times the upper limit of the normal range) and coagulation (international normalized ratio <2.3) function.

Exclusion Criteria:

* Exclusion criteria included a history of treatment with immune checkpoint inhibitors, allergies to immunetherapeutics, systemic immunosuppressive therapy, and ongoing or active infection, or an active autoimmune disease.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Adverse events | 6-8 weeks
  Safety evaluation was done continuously during ICIs treatment and up to 30 days after the last dose by using the Common Terminology Criteria for Adverse Events (CTCAE; version 4.03). Complications related to ablation procedure were assessed peri-operation period and reported according to the standardized Society of Interventional Radiology grading system.
Response | 6-8 weeks
  Efficacy included objective response (includes complete and partial response), duration of response, and disease control (Includes complete and partial response, stable disease and atypical progression for at least 3 months).

SECONDARY OUTCOMES:
Time to tumor progression | 3-4 months
  time from first dose of ICIs drug until the first typical progression of disease
Progression-free survival | 3-4 months
  time from first day of ICIs treatment to first typical disease progression, or death, which occurred earlier
Overall survival | 3-4 months
  time from first study treatment to death of any cause

CONTACTS AND LOCATIONS:
Overall Officials: Ming Zhao, MD, Ph.D, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lyu N, Kong Y, Li X, Mu L, Deng H, Chen H, He M, Lai J, Li J, Tang H, Lin Y, Zhao M. Ablation Reboots the Response in Advanced Hepatocellular Carcinoma With Stable or Atypical Response During PD-1 Therapy: A Proof-of-Concept Study. Front Oncol. 2020 Oct 9;10:580241. doi: 10.3389/fonc.2020.580241. eCollection 2020. PMID 33163408